CLINICAL TRIAL: NCT00224952
Title: The Role of Drug Metabolizing Enzymes in the Pathogenesis Adverse Drug Reactions in Children
Brief Title: Pathogenesis of Adverse Drug Reactions
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Utah (Other); University of Louisville (Other)
Responsible Party: Principal Investigator, Steve Leeder, Pharm.D; Ph.D, Children's Mercy Hospital Kansas City
Other Study IDs: PPRU 10606; NIH Grant HD044239
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Seizures
Keywords: seizures; Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Urine Specimen Collection; Carbamazepine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine DNA (source: blood or saliva)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving Carbamazepine or Valproic Acid
  Interventions: Other: No intervention; Urine Collection

INTERVENTIONS:
Other: No intervention; Urine Collection — Urine collected from children receiving carbamazepine or valproic acid as part of their clinical management
  Other Names: carbamazepine: Tegretol; valproic acid: Depakote

SUMMARY:
The purpose of the study is to examine the individual metabolic profiles of pediatric patients receiving carbamazepine or valproate therapy, in an attempt to determine identities of the reactive metabolites or, alternatively, the identities of those metabolites that serve as potential precursors to reactive species.

DETAILED DESCRIPTION:
Adverse drug reactions can be broadly defined as any undesirable response associated with therapeutic drug use. A simple and clinically useful classification is to divide adverse events into those that are dose-dependent and largely predictable from the known pharmacologic properties of the compound in question, and those that are dependent on characteristics unique to susceptible individuals, or idiosyncratic in nature.

The long term objective of this research is to characterize the mechanisms responsible for the pathogenesis of idiosyncratic hypersensitivity reactions in children, particularly those involving carbamazepine and other aromatic anticonvulsants.

The study is divided into two phases. Phase 1 of the study involves collecting urine from 50 patients taking CBZ therapeutically. Participants will be asked to provide a spot urine sample during routine health visits. The urine will be analyzed for the presence of CBZ and its metabolites. In Phase 2 of the study, urine will be collected from patients taking either CBZ or VPA therapeutically. If blood samples are drawn from these patients for medical purposes not related to this study the residual blood sample will be recovered before it is discarded for use in genotyping analysis. Participants will be asked to provide a urine sample covering one complete dosing interval of CBZ or VPA (preferably overnight). Patients will also be followed longitudinally, with urine collections at each clinic visit over at least a two year period.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients of both genders between 1 and 16 years of age receiving CBZ or VPA mono-therapy will be recruited for this study. Additionally, for those patients who are receiving drugs other than CBZ or VPA to control their seizures, if CBZ or VPA are subsequently added to their treatment regimen, then these patients will also be recruited for this study.

Exclusion Criteria:

* None

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients of both genders between 1 and 16 years of age receiving carbamazepine (CBZ) or valproic acid (VPA) as monotherapy or polytherapy
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2002-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Steven Leeder, Pharm.D., Ph.D.,, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (3):
- United States (3):
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Mercy Hospital, Kansas City, Missouri
  - Primary Children's Hospital, Pediatric Neurology, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbamazepine Phase 1; Carbamazepine Phase 2: No intervention; Urine Collection: Urine collected from children receiving carbamazepine as part of their clinical management
- Valporic Acid Phase 2: No intervention; Urine Collection: Urine collected from children receiving valproic acid as part of their clinical management
Period: Overall Study
Arm/Group | Carbamazepine Phase 1 | Carbamazepine Phase 2 | Valporic Acid Phase 2
Started | 53 | 87 | 134
Completed | 53 | 87 | 134
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbamazepine Phase 1 | Carbamazepine Phase 2 | Valporic Acid Phase 2 | Total
Number analyzed (Participants) | 53 | 87 | 134 | 274
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.8 (4.6) | 11.0 (4.0) | 10.2 (4.1) | 10.38 (4.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 43 | 56 | 117
  Male | 35 | 44 | 78 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7 | 14
  Not Hispanic or Latino | 52 | 81 | 127 | 260
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 14 | 18
  White | 47 | 80 | 111 | 238
  More than one race | 2 | 5 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Drug (Valproic Acid or Carbamazepine) Metabolite Profiles in Urine
Description: 1. To examine the individual metabolic profiles of pediatric patients receiving carbamazepine or valproate therapy, in an attempt to determine the identities of the reactive metabolites or, alternatively, the identities of those metabolites that serve as potential precursors to reactive species (e.g., through conjugation with detoxifying compounds such as glutathione).
Time Frame: urine samples (overnight collections) collected longitudinally through study completion for time frame ranging from 2-5 years
Population: Carbamazepine detoxification product (MTHIS) was only measured in the Carbamazepine Phase I and 2 arms. Valproic Acid (NAC) detoxification products were only measured in the Valproic Acid Phase 2 arm. Units of measure for all analytes are nmol per mg creatinine.
Measure: Mean (Standard Deviation); unit: nmol per mg creatinine
Groups:
- Valproic Acid Phase 2: No intervention; Urine Collection: Urine collected from children receiving valproic acid as part of their clinical management
Arm/Group | Carbamazepine Phase 1 | Carbamazepine Phase 2 | Valproic Acid Phase 2
Number analyzed (Participants) | 53 | 87 | 134
nmol per mg creatinine
  4-Methylthio-2-hydroxyiminostilbene: number analyzed (Participants) | 53 | 87 | 0
  4-Methylthio-2-hydroxyiminostilbene | 15.2 (28.1) | 13.1 (11.5) |
  5-N-acetylcysteine-3-ene VPA isomers: number analyzed (Participants) | 0 | 0 | 134
  5-N-acetylcysteine-3-ene VPA isomers |  |  | 1.15 (1.20)
  5-N-acetylcysteine-2-ene VPA: number analyzed (Participants) | 0 | 0 | 134
  5-N-acetylcysteine-2-ene VPA |  |  | 2.13 (1.68)
  Total N-acetylcysteine conjugates: number analyzed (Participants) | 0 | 0 | 134
  Total N-acetylcysteine conjugates |  |  | 5.88 (5.17)

2. Secondary Outcome: Age-related Changes in Bioactivation
Description: 2. To determine if age-related differences exist regarding the ability of pediatric patients to bioactivate carbamazepine or valproate to reactive metabolites. Data provided below reflect the slope of the least squares regression.
Time Frame: as for outcome 1
Population: Change in Carbamazepine detoxification as a function of age is determined only in patients in the Carbamazepine Phase 2 arm. Changes in Valproic Acid detoxification as a function of age are determined only in patients in the Valproic Acid Phase 2 arm.
Measure: Number; unit: years^(-1)
Arm/Group | Carbamazepine Phase 1 | Carbamazepine Phase 2 | Valporic Acid Phase 2
Number analyzed (Participants) | 0 | 87 | 134
years^(-1)
  4-Methylthio-2-hydroxyiminostilbene: number analyzed (Participants) | 0 | 87 | 0
  4-Methylthio-2-hydroxyiminostilbene |  | -0.8876 |
  Log (4-Methylthio-2-hydroxyiminostilbene): number analyzed (Participants) | 0 | 87 | 0
  Log (4-Methylthio-2-hydroxyiminostilbene) |  | -0.0244 |
  Fractional Recovery MTHIS: number analyzed (Participants) | 0 | 87 | 0
  Fractional Recovery MTHIS |  | -0.00033 |
  Log (Fractional Recovery MTHIS): number analyzed (Participants) | 0 | 87 | 0
  Log (Fractional Recovery MTHIS) |  | -00122 |
  Log (5-N-acetylcysteine-3-ene VPA isomers): number analyzed (Participants) | 0 | 0 | 134
  Log (5-N-acetylcysteine-3-ene VPA isomers) |  |  | -0.0295
  Log (5-N-acetylcysteine-2-ene VPA): number analyzed (Participants) | 0 | 0 | 134
  Log (5-N-acetylcysteine-2-ene VPA) |  |  | -0.0250
  Total N-acetylcysteine conjugates: number analyzed (Participants) | 0 | 0 | 134
  Total N-acetylcysteine conjugates |  |  | -0.0296
  Log (Fractional Recovery NAC-3-ene VPA isomers): number analyzed (Participants) | 0 | 0 | 134
  Log (Fractional Recovery NAC-3-ene VPA isomers) |  |  | -0.005155
  Log (Fractional Recovery NAC-2-ene VPA): number analyzed (Participants) | 0 | 0 | 134
  Log (Fractional Recovery NAC-2-ene VPA) |  |  | -0.000698
  Log (Fractional Recovery Total NAC conjugates): number analyzed (Participants) | 0 | 0 | 134
  Log (Fractional Recovery Total NAC conjugates) |  |  | -0.005272
Statistical Analysis 1: Comparison: Carbamazepine Phase 2; Least squares linear regression evaluating fractional analyte recovery (4-Methylthio-2-hydroxyiminostilbene) as a function of age; Test type: Other; p = 0.004, Regression, Linear
Statistical Analysis 2: Comparison: Carbamazepine Phase 2; Least squares linear regression evaluating fractional analyte recovery (Log (4-Methylthio-2-hydroxyiminostilbene) as a function of age; Test type: Other; p = 0.032, Regression, Linear
Statistical Analysis 3: Comparison: Carbamazepine Phase 2; Least squares linear regression evaluating fractional analyte recovery (Fractional Recovery (MTHIS)) as a function of age; Test type: Other; p = 0.018, Regression, Linear
Statistical Analysis 4: Comparison: Carbamazepine Phase 2; Least squares linear regression evaluating fractional analyte recovery (Log (Fractional Recovery MTHIS)) as a function of age; Test type: Other; p = 0.033, Regression, Linear
Statistical Analysis 5: Comparison: Valporic Acid Phase 2; Least squares linear regression evaluating fractional analyte recovery (Log (5-N-acetylcysteine-3-ene VPA isomers)) as a function of age; Test type: Other; p = 0.0004, Regression, Linear
Statistical Analysis 6: Comparison: Valporic Acid Phase 2; Least squares linear regression evaluating fractional analyte recovery (Log (5-N-acetylcysteine-2-ene VPA) ) as a function of age; Test type: Other; p = 0.0003, Regression, Linear
Statistical Analysis 7: Comparison: Valporic Acid Phase 2; Least squares linear regression evaluating fractional analyte recovery (Total N-acetylcysteine conjugates) as a function of age; Test type: Other; p < 0.0001, Regression, Linear
Statistical Analysis 8: Comparison: Valporic Acid Phase 2; Least squares linear regression evaluating fractional analyte recovery (Log (Fractional Recovery NAC-3-ene VPA isomers)) as a function of age; Test type: Other; p = 0.522, Regression, Linear
Statistical Analysis 9: Comparison: Valporic Acid Phase 2; Least squares linear regression evaluating fractional analyte recovery (Log (Fractional Recovery NAC-2-ene VPA) ) as a function of age; Test type: Other; p = 0.925, Regression, Linear
Statistical Analysis 10: Comparison: Valporic Acid Phase 2; Least squares linear regression evaluating fractional analyte recovery (Log (Fractional Recovery Total NAC conjugates) as a function of age; Test type: Other; p = 0.469, Regression, Linear

ADVERSE EVENTS:
Description: This was an observational study with no interventions. The study posed no significant risks to participants thus explaining 0 participants at risk.
Arm/Group | Carbamazepine Phase 1 | Carbamazepine Phase 2 | Valporic Acid Phase 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes